CLINICAL TRIAL: NCT01666275
Title: The Metabolomics of Anaphylaxis
Status: Withdrawn | Type: Observational
Why Stopped: We are closing the study because of lack of enrollment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aleena Banerji, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2012P000448
Record Dates: First submitted 2012-08-07; First posted 2012-08-16 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Patients With AERD Undergoing Aspirin Desensitization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We retain and freeze the plasma from blood after spinning down whole-blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspirin desensitization: This group of patients has AERD (aspirin exacerbated respiratory disease) and is undergoing aspirin desensitization.

SUMMARY:
Metabolomics is the study of metabolic pathways and the unique biochemical molecules which result from the regulatory response to physiological stressors, disease processes, or drug therapy. By measuring changes in metabolite concentrations, the range of biochemical effects and therapeutic intervention can be determined.

Aspirin exacerbated respiratory disease (AERD) is a chronic inflammatory disease characterized by chronic rhinosinusitis, nasal polyposis, asthma, and airway reactivity to aspirin and/or other nonsteroidal anti-inflammatory drugs (NSAIDs). This reaction to aspirin during challenge/desensitization is equivalent to an allergic drug reaction however we are able to evaluate these specific reactions in a controlled, clinical environment. This population of patients undergoing aspirin desensitization is ideal for studying metabolomics as serial blood sampling can be performed in patients before, during a reaction, and after aspirin desensitization, thereby allowing each patient to serve as his or her own biological control. The investigator hopes that this study of metabolomics will allow for better methods of identifying anaphylaxis in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-75 with a history of aspirin anaphylaxis or a history of hypersensitivity reaction to aspirin and referred for a clinically indicated outpatient or inpatient aspirin desensitization procedure for AERD.

Exclusion Criteria:

* Pregnancy/breastfeeding, possibility of poor compliance, unwilling to undergo aspirin desensitization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 18-75, history of an allergic reaction to aspirin and referred for a clinically indicated outpatient or inpatient aspirin desensitization procedure for aspirin exacerbated respiratory disease (AERD)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Change in metabolic profile of blood serum metabolites from Baseline to 1 week post-desensitization | before start of aspirin desensitization, 2 hours into desensitization, at time of reaction(s) - an expected average of 6 hours into desensitization, 1 week post-desensitization
  Metabolic profiling will be done on specific blood serum metabolites including lipid mediators, amino acids, and leukotrienes.

CONTACTS AND LOCATIONS:
Overall Officials: Aleena S Banerji, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Allergy Associates, Boston, Massachusetts, United States